CLINICAL TRIAL: NCT04477473
Title: Perceived Impact of the COVID-19 Pandemic on Medical Management and Symptoms in a High Risk Group: Patients Under Long Term Noninvasive Ventilation for Chronic Hypercapnic Respiratory Failure in Geneva. An Observational Monocentric Study
Brief Title: Perceived Impact of the COVID-19 Pandemic on Medical Management and Symptoms in a High Risk Group
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jean-Paul Janssens, Professor, University Hospital, Geneva
Other Study IDs: 2020-01509
Record Dates: First submitted 2020-07-17; First posted 2020-07-20 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: COVID-19 Pandemic; Vulnerable Subjects; Long-term Non-invasive Ventilation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vulnerable subjects: Patients under long-term non-invasive ventilation (respiratory support) at home for chronic respiratory failure
  Interventions: Other: Questionnaire-based observational study

INTERVENTIONS:
Other: Questionnaire-based observational study — Questionnaire focusing on practical health care issues regarding respiratory support, health status and perception of the COVID-19 issue:
  * Symptom score (related to noninvasive ventilation: NIV)
  * Thymic disturbances (score of anxiety and depression)
  * Compliance to treatment (assessed via tele-monitoring: routine procedure)

SUMMARY:
The Swiss population underwent a period of confinement related to the COVID-19 pandemic (March 16 to May 11, 2020) decided by the Swiss Federal Government. Among the Swiss population, certain groups were identified as vulnerable subjects by the Federal Office of Public Health. This study focuses on the perceived impact of this period on health care and health status in a specific vulnerable group: patients under long term noninvasive ventilation (respiratory support) at home for chronic respiratory failure.

DETAILED DESCRIPTION:
The Swiss population underwent a period of confinement related to the COVID-19 pandemic (March 16 to May 11, 2020) decided by the Swiss Federal Government. Among the Swiss population, certain groups were identified as vulnerable subjects by the Federal Office of Public Health. This study focuses on the perceived impact of this period on health care and health status in a specific vulnerable group: patients under long term noninvasive ventilation (respiratory support) at home for chronic respiratory failure.

The objective is to determine, in a specific vulnerable group, how the confinement related to the COVID-19 pandemic affected health care and health status, as perceived by the patients.

The primary outcome is a questionnaire focusing on practical health care issues regarding respiratory support, health status and perception of the COVID-19 issue:

* Symptom score (related to noninvasive ventilation: NIV)
* Thymic disturbances (score of anxiety and depression)
* Compliance to treatment (assessed via tele-monitoring: routine procedure)

It is a non-interventional questionnaire-based observational study of patients followed by the Division of Pulmonology of Geneva University Hospitals with home NIV, aged above 18 years of age and in a stable clinical condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed by the Division of Pulmonology of Geneva University Hospitals with home NIV
* Aged above 18 years of age
* Stable clinical condition

Exclusion Criteria:

* Age below 18 years of age
* Unwillingness to participate
* Unstable clinical condition

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population chosen (patients with chronic hypercapnic respiratory failure treated by noninvasive ventilation) is:
  * One of the main focuses of interest of our research group, for close to 30 years
  * One of our main clinical activities in our outpatient pulmonary division
  * An interesting group because, although these subjects must be considered as vulnerable in case of COVID-19, they have - albeit for COPD - a prognosis of several years of survival
  * A group for which the findings of our study can be rapidly translated into adapting clinical practice and management
  * An interesting group because although they are often very limited in their activities of daily life (ADL), they are also very resilient, with remarkable coping strategies
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Questionnaire | 2 months
  Questionnaire focusing on practical health care issues regarding respiratory support, health status and perception of the COVID-19 issue:
  * Symptom score (related to noninvasive ventilation: NIV): S3-NIV (non-invasive ventilation), score ranging from 0 to 10, the lowest possible score (0) corresponds to the highest impact of disease and treatment, the highest possible score (10) corresponds to the lowest impact of disease and treatment.
  * Thymic disturbances (score of anxiety and depression): HADS (Hospital Anxiety and Depression Scale), score ranging from 0 to 21, 0-7 = normal, 8-10 borderline abnormal, 11-21 =abnormal
  * COVID confinement questionnaire: de novo questionnaire, Minimal Clinically Important Differences (MCID) unknown

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Janssens, M.D, Principal Investigator — University Hospital, Geneva
Locations (1):
- Centre antituberculeux; Geneva University Hospital, Geneva, Geneva 14, Switzerland